CLINICAL TRIAL: NCT02426632
Title: A Phase 1, Double-blind, Randomized, Trial to Evaluate the Taste Profile of Different JNJ-53718678 Oral Liquid Formulations in Healthy Subjects
Brief Title: Study to Evaluate Taste Profile of Different JNJ-53718678 Oral Liquid Formulations in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Sciences Ireland UC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: CR106726; 53718678RSV1003 (Other: Janssen Sciences Ireland UC); 2014-005157-39 (EudraCT Number)
Record Dates: First submitted 2015-04-22; First posted 2015-04-27 (Estimated); Last update posted 2018-05-15 (Actual); Status verified 2018-05

CONDITIONS: Healthy
Keywords: Healthy; JNJ-53718678
MeSH Terms: interventions — JNJ-53718678; D-Worm; Granuflex E

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No

ARMS (12):
- Session 1: Sequence 1 (Experimental): Participants will sequentially receive 5 milliliter of each 6 JNJ-53718678 formulations (ABCDEF) in a random order, at a dosing interval of 1-2 hours.
  Interventions: Drug: Formulation A; Drug: Formulation B; Drug: Formulation C; Drug: Formulation D; Drug: Formulation E; Drug: Formulation F
- Session 1: Sequence 2 (Experimental): Participants will sequentially receive 5 milliliter of each 6 JNJ-53718678 formulations (ABCDEF) in a random order, at a dosing interval of 1-2 hours.
  Interventions: Drug: Formulation A; Drug: Formulation B; Drug: Formulation C; Drug: Formulation D; Drug: Formulation E; Drug: Formulation F
- Session 1: Sequence 3 (Experimental): Participants will sequentially receive 5 milliliter of each 6 JNJ-53718678 formulations (ABCDEF) in a random order, at a dosing interval of 1-2 hours.
  Interventions: Drug: Formulation A; Drug: Formulation B; Drug: Formulation C; Drug: Formulation D; Drug: Formulation E; Drug: Formulation F
- Session 1: Sequence 4 (Experimental): Participants will sequentially receive 5 milliliter of each 6 JNJ-53718678 formulations (ABCDEF) in a random order, at a dosing interval of 1-2 hours.
  Interventions: Drug: Formulation A; Drug: Formulation B; Drug: Formulation C; Drug: Formulation D; Drug: Formulation E; Drug: Formulation F
- Session 1: Sequence 5 (Experimental): Participants will sequentially receive 5 milliliter of each 6 JNJ-53718678 formulations (ABCDEF) in a random order, at a dosing interval of 1-2 hours.
  Interventions: Drug: Formulation A; Drug: Formulation B; Drug: Formulation C; Drug: Formulation D; Drug: Formulation E; Drug: Formulation F
- Session 1: Sequence 6 (Experimental): Participants will sequentially receive 5 milliliter of each 6 JNJ-53718678 formulations (ABCDEF) in a random order, at a dosing interval of 1-2 hours.
  Interventions: Drug: Formulation A; Drug: Formulation B; Drug: Formulation C; Drug: Formulation D; Drug: Formulation E; Drug: Formulation F
- Session 2: Sequence 7 (Experimental): Participants will receive two best scoring formulations from Session 1 with a varying concentration of sucralose (M1M2M3N1N2N3) sequentially in a random order, at a dosing interval of 1-2 hours.
  Interventions: Drug: Formulation M1; Drug: Formulation M2; Drug: Formulation M3; Drug: Formulation N1; Drug: Formulation N2; Drug: Formulation N3
- Session 2: Sequence 8 (Experimental): Participants will receive two best scoring formulations from Session 1 with a varying concentration of sucralose (M1M2M3N1N2N3) sequentially in a random order, at a dosing interval of 1-2 hours.
  Interventions: Drug: Formulation M1; Drug: Formulation M2; Drug: Formulation M3; Drug: Formulation N1; Drug: Formulation N2; Drug: Formulation N3
- Session 2: Sequence 9 (Experimental): Participants will receive two best scoring formulations from Session 1 with a varying concentration of sucralose (M1M2M3N1N2N3) sequentially in a random order, at a dosing interval of 1-2 hours.
  Interventions: Drug: Formulation M1; Drug: Formulation M2; Drug: Formulation M3; Drug: Formulation N1; Drug: Formulation N2; Drug: Formulation N3
- Session 2: Sequence 10 (Experimental): Participants will receive two best scoring formulations from Session 1 with a varying concentration of sucralose (M1M2M3N1N2N3) sequentially in a random order, at a dosing interval of 1-2 hours.
  Interventions: Drug: Formulation M1; Drug: Formulation M2; Drug: Formulation M3; Drug: Formulation N1; Drug: Formulation N2; Drug: Formulation N3
- Session 2: Sequence 11 (Experimental): Participants will receive two best scoring formulations from Session 1 with a varying concentration of sucralose (M1M2M3N1N2N3) sequentially in a random order, at a dosing interval of 1-2 hours.
  Interventions: Drug: Formulation M1; Drug: Formulation M2; Drug: Formulation M3; Drug: Formulation N1; Drug: Formulation N2; Drug: Formulation N3
- Session 2: Sequence 12 (Experimental): Participants will receive two best scoring formulations from Session 1 with a varying concentration of sucralose (M1M2M3N1N2N3) sequentially in a random order, at a dosing interval of 1-2 hours.
  Interventions: Drug: Formulation M1; Drug: Formulation M2; Drug: Formulation M3; Drug: Formulation N1; Drug: Formulation N2; Drug: Formulation N3

INTERVENTIONS:
Drug: Formulation A — Reference formulation, 10 milligram/milliliter (mg/mL)oral solution without sweetener/flavor.
  Other Names: JNJ-53718678
  Arms: Session 1: Sequence 1; Session 1: Sequence 2; Session 1: Sequence 3; Session 1: Sequence 4; Session 1: Sequence 5; Session 1: Sequence 6
Drug: Formulation B — 10 mg/mL oral solution containing 2 mg/mL sucralose, masking flavor and orange flavor.
  Other Names: JNJ-53718678
  Arms: Session 1: Sequence 1; Session 1: Sequence 2; Session 1: Sequence 3; Session 1: Sequence 4; Session 1: Sequence 5; Session 1: Sequence 6
Drug: Formulation C — 10 mg/mL oral solution containing 10 mg/mL sucralose.
  Other Names: JNJ-53718678
  Arms: Session 1: Sequence 1; Session 1: Sequence 2; Session 1: Sequence 3; Session 1: Sequence 4; Session 1: Sequence 5; Session 1: Sequence 6
Drug: Formulation D — 10 mg/mL oral solution containing 2 mg/mL sucralose and raspberry flavor.
  Other Names: JNJ-53718678
  Arms: Session 1: Sequence 1; Session 1: Sequence 2; Session 1: Sequence 3; Session 1: Sequence 4; Session 1: Sequence 5; Session 1: Sequence 6
Drug: Formulation E — 10 mg/mL oral solution containing 2 mg/mL sucralose and strawberry flavor.
  Other Names: JNJ-53718678
  Arms: Session 1: Sequence 1; Session 1: Sequence 2; Session 1: Sequence 3; Session 1: Sequence 4; Session 1: Sequence 5; Session 1: Sequence 6
Drug: Formulation F — 10 mg/mL oral solution containing 2 mg/mL sucralose and orange flavor.
  Other Names: JNJ-53718678
  Arms: Session 1: Sequence 1; Session 1: Sequence 2; Session 1: Sequence 3; Session 1: Sequence 4; Session 1: Sequence 5; Session 1: Sequence 6
Drug: Formulation M1 — Best scoring formulation from Session 1 with a varying concentration of sucralose (maximum 10 mg/mL).
  Other Names: JNJ-53718678
  Arms: Session 2: Sequence 10; Session 2: Sequence 11; Session 2: Sequence 12; Session 2: Sequence 7; Session 2: Sequence 8; Session 2: Sequence 9
Drug: Formulation M2 — Best scoring formulation from Session 1 with a varying concentration of sucralose (maximum 10 mg/mL).
  Other Names: JNJ-53718678
  Arms: Session 2: Sequence 10; Session 2: Sequence 11; Session 2: Sequence 12; Session 2: Sequence 7; Session 2: Sequence 8; Session 2: Sequence 9
Drug: Formulation M3 — Best scoring formulation from Session 1 with a varying concentration of sucralose (maximum 10 mg/mL).
  Other Names: JNJ-53718678
  Arms: Session 2: Sequence 10; Session 2: Sequence 11; Session 2: Sequence 12; Session 2: Sequence 7; Session 2: Sequence 8; Session 2: Sequence 9
Drug: Formulation N1 — Second best scoring formulation from Session 1 with a varying concentration of sucralose (maximum 10 mg/mL).
  Other Names: JNJ-53718678
  Arms: Session 2: Sequence 10; Session 2: Sequence 11; Session 2: Sequence 12; Session 2: Sequence 7; Session 2: Sequence 8; Session 2: Sequence 9
Drug: Formulation N2 — Second best scoring formulation from Session 1 with a varying concentration of sucralose (maximum 10 mg/mL).
  Other Names: JNJ-53718678
  Arms: Session 2: Sequence 10; Session 2: Sequence 11; Session 2: Sequence 12; Session 2: Sequence 7; Session 2: Sequence 8; Session 2: Sequence 9
Drug: Formulation N3 — Second best scoring formulation from Session 1 with a varying concentration of sucralose (maximum 10 mg/mL).
  Other Names: JNJ-53718678
  Arms: Session 2: Sequence 10; Session 2: Sequence 11; Session 2: Sequence 12; Session 2: Sequence 7; Session 2: Sequence 8; Session 2: Sequence 9

SUMMARY:
The primary objective is to evaluate in a double-blinded (neither physician nor participant knows the treatment that the participant receives), fashion the taste of different JNJ-53718678 oral liquid formulations as compared to the reference formulation (JNJ-53718678, 10 milligram/milliliter oral solution without sweetener/flavor).

DETAILED DESCRIPTION:
This is a Phase 1, double-blind, randomized (participants taste the same groups of drugs [formulations] but in random order), single-center trial in healthy adult participants. The study will include 2 Sessions of 1 day, 1) Session 1, in which participants will receive 6 JNJ-53718678 oral solutions (1 reference and 5 different formulations) sequentially in a randomized order, Scoring of the taste will be done via a questionnaire designed for this purpose; 2) Session 2, within approximately a timeframe of 7 to 14 days after completion of Session 1, participants will taste 2 best scoring tastes coming out of Session 1. The study will consist of a screening phase of approximately 2 weeks, treatment phase of approximately 2 weeks and a post-treatment follow-up phase of 10 days after completion of the last Session. The total study duration for each participant will be approximately 6 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Female participants of childbearing potential should have a urine pregnancy test at screening which should be negative
* Participants must be non-smokers and/or have not used chewing tobacco for at least one month prior to screening
* Participants must be willing/able to adhere to the prohibitions and restrictions specified in the protocol and study procedures
* Participants must be able to taste and smell normally, to their own opinion, at all times throughout the study duration. Participants who have an impaired sense of taste and/or smell due to any conditions like common cold or sinusitis are not eligible to take part or to continue to study
* Participants must agree to use an adequate method of contraception

Exclusion Criteria:

* Participant has a mouth pathology including, but not limited to, pain, ulcer, edema, mucosal erosion, and/or (dental) abscesses, or receives treatment for oral pathologies or oral treatment for any disease
* Participant has a history of any illness that, in the opinion of the Investigator, might confound the results of the study or pose an additional risk in administering study drug to the participant or that could prevent, limit or confound the protocol specified assessments. This may include but is not limited to renal dysfunction, significant cardiac, vascular, pulmonary, gastrointestinal (such as significant diarrhea, gastric stasis, or constipation that in the Investigator's opinion could influence drug absorption or bioavailability), endocrine, neurologic, hematologic, rheumatologic, psychiatric, neoplastic, or metabolic disturbances
* Participants with a history of clinically significant allergies, hypersensitivity, or intolerance to drugs such as, but not limited to, sulfonamides and penicillins, drug allergy witnessed in previous studies with experimental drugs, or to JNJ-53718678 or its excipients
* Participants with a history or evidence of use of alcohol, barbiturates, amphetamines, recreational or narcotic drug use within the past 3 months, which in the Investigator's opinion would compromise participant's safety and/or compliance with the study procedures
* Participants having received an investigational drug (including investigational vaccines) or used an invasive investigational device within 3 months before the planned first dose of study drugs or is currently enrolled in an investigational study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2015-03-04 (Actual); Primary Completion 2015-04-24 (Actual); Study Completion 2015-04-24 (Actual)

PRIMARY OUTCOMES:
Acceptability Score | up to 12 hour post-administration of study drug
  Formulations will be assessed using Acceptability Questionnaire, which evaluates sweetness, bitterness, aroma type, aroma strength, smell and overall acceptability using visual analogue scales (VAS) with range from 0 (super bad) to 100 (super good).

SECONDARY OUTCOMES:
Number of Participants with Local and Systemic adverse Events | Screening up to end of Study (Week 6)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Sciences Ireland UC Clinical Trial, Study Director — Janssen Sciences Ireland UC
Locations (1):
- Nottingham, United Kingdom